CLINICAL TRIAL: NCT04633837
Title: A Prospective Double Blinded Randomized Controlled Trial Examining the Effectiveness of a Connective Tissue Matrix Implant in Reducing Post-operative Pain and Narcotic Use in Patients Under 55yo After Outpatient Arthroscopic Shoulder Surgery
Brief Title: Examining the Effectiveness of a Connective Tissue Matrix Implant in Reducing Post-operative Pain and Narcotic After Outpatient Arthroscopic Shoulder Surgery
Acronym: ECM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Left employment with job and study site
Sponsor: Brian Badman (Other)
Collaborators: CTM Biomedical (Industry)
Responsible Party: Sponsor-Investigator, Brian Badman, Orthopedic Surgeon, Indiana University
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1294348
Record Dates: First submitted 2020-11-01; First posted 2020-11-18 (Actual); Results first posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Arthroscopic Shoulder Surgery; Pain, Postoperative
Keywords: extracellular matrix implant
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: The extracellular matrix implant injection is the intervention in this study. One group of patients undergoing arthroscopic shoulder surgery will receive 2cc of the injectable implant placed into the glenohumeral joint space at completion of the rotator cuff repair and the other group will not.
Who Masked: Participant, Care Provider, Investigator
Masking Description: This is a double-blinded study, thus, neither the surgeon nor the patient will know if the extracellular matrix injection was given. A total of 70 envelopes will be made with 35 containing a card designating "treatment" and 35 designating "control". Envelopes will be randomly opened at completion of the surgery and if the treatment group is selected the patient will be administered the injectable extracellular matrix graft. Dr. Badman will place a 22 gauge needle transtendon into the glenohumeral joint space and will then exit the room prior to the envelope being opened. If the treatment group is selected, his physician assistant will administer the injection. If the control group is selected, the needle will be removed and no injection will be given.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group 1 Control (No Intervention): Group 1 will undergo standard arthroscopic shoulder surgery without the ECM injection.
- Group 2: ECM Injectable graft (Active Comparator): Group 2 will undergo arthroscopic shoulder surgery and receive 2cc of the injectable extracellular matrix injection placed into the glenohumeral joint space via a transtendon approach at the end of the surgery
  Interventions: Device: Extracellular Matrix Graft Injectable Implant

INTERVENTIONS:
Device: Extracellular Matrix Graft Injectable Implant — The extracellular matrix injectable implant will serve as the intervention in this study.
  Other Names: CTM graft
  Arms: Group 2: ECM Injectable graft

SUMMARY:
This document is a protocol for a human research study. This study is to be conducted according to United States standards of Good Clinical Practice in accordance with applicable Federal regulations and institutional research policies and procedures.

Extracellular matrix grafts have been used to help with postoperative inflammation.

DETAILED DESCRIPTION:
Shoulder surgery has evolved over the past decade with many procedures now done on an outpatient basis. Multimodal pain management strategies and regional anesthesia have greatly contributed to this transition and newer strategies continue to evolve. Uncontrolled pain can often lead to readmissions, prolonged hospital or ambulatory stays and an overall negative patient experience. Despite improvements in regional anesthetic technique and newer longer acting medicines such as liposomal bupivacaine, the duration of pain relief is often only over the course of 72 hours postoperatively. Post-operative pain beyond 72 hours is largely inflammatory in nature. As such, biologic approaches to reduce surgical tissue damage-induced inflammation is an attractive therapeutic addition to surgical procedures. These approaches are especially relevant in light of the current opioid epidemic plaguing the United States.

Flowable, placental-derived connective tissue matrix (pECM) is a potential option to supplement damaged tissue prone to inflammation as it introduces nascent, hydrated components of the inflammatory phase, including structural proteins and growth factors, which allow for efficient repair. Derived from relatively immune-privileged tissue, placental-derived pECM elicits little or no immune response in recipients. They have been shown to greatly reduce inflammatory cell influx and inflammatory cytokines present in dermal and mucosal surgical sites post-operatively. Moreover, placental-derived pECM reduces expression of prostaglandin E2, a potent pain mediator, in vitro. In the orthopedic space, ECM has been used effectively to reduce pain following spinal fusion and for treatment of knee arthritis. Taken together, biologic therapies directed at modulating inflammation and associated pain is an increasing area of interest with far reaching implications.

The purpose of the current study is to prospectively analyze two groups of patients treated for arthroscopic shoulder surgery with and without a flowable pECM to determine if a significant reduction in pain and opioid consumption as measured in morphine equivalent units is demonstrated within the first 6 weeks of surgery. Furthermore, patients will be compared in regard to early range of motion and patient reported outcomes to determine if a difference is present when the ECM is utilized within the first 6 months of surgery. This is the first double blinded prospective series in the shoulder literature to date looking at a pECM graft for pain reduction and improved range of motion perioperatively.

Study Objectives

Utilizing a prospective randomized controlled trial, the aim of this study is to assess modulation of post-operative pain and narcotic use when a placental-derived extracellular matrix is injected into the bed of the repair following outpatient arthroscopic shoulder surgery. Furthermore, this study aims to determine if the addition of pECM influences patient reported outcomes and influences early postoperative range of motion.

Primary Aims & Objective

Aim 1a: To assess post-operative narcotic consumption (measured in morphine equivalent units) between patients treated with flowable placental-derived pECM compared to those patients undergoing arthroscopic shoulder surgery.

Hypothesis: Narcotic consumption (measured in morphine equivalent units) will be reduced in patients treated with an extracullar matrix graft as compared to those patients undergoing rotator cuff surgery without.

Objective: Utilizing a prospective randomized controlled trial, narcotic use will be measured for 24-hour increments for a total of 7 post-operative days (PODs) then once on POD 14, 21, 28, and 42. . Consumption will be measured by the number of tablets ingested and converted to morphine equivalent units and compared between the two treatment groups.

Aim 1b: To determine if flowable placental-derived pECM decreases patient-reported post-operative VAS pain in patients undergoing outpatient rotator cuff surgery

Hypothesis: There will be a decrease in VAS pain for up to 6 weeks post-operatively among participants who receive pECM, as compared to the control group (no pECM).

Objective: Utilizing a prospective randomized controlled trial, post-operative patient-reported VAS pain (on a scale of 0-10) will be collected 1 times per day (every 24 hours) for 7 post-operative days (PODs); then an average score collected on POD 14, POD 21, POD 28, and POD 42. Scores will be averaged and compared between the two treatment groups for the first 7 days, 2 week, 3rd week, 4th week and 6th week postoperatively.

Secondary Aims & Objectives

Aim 2a: To assess patient-reported outcomes and early range of motion (measured in morphine equivalents) in patients treated with flowable placental-derived pECM compared to patients injected with saline control.

Hypothesis: There will be improved patient reported outcomes and early range of motion measured at 6 weeks and 3 months and 6 months postoperatively in patients receiving and extracellular matrix injection following outpatient arthroscopic shoulder surgery.

Objective: Utilizing a prospective randomized controlled trial, patient reported outcomes as measured by American Shoulder and Elbow Score, Simple Shoulder Test and SANE scores and range of motion (External rotation, internal rotation and forward flexion) will be collected preoperatively and at 2 weeks (external rotation), 6 weeks (all)) , 3 months (all) and 6 months (all) postoperatively. Scores and range of motion measurements will be averaged and compared for differences between the two groups.

Study Design

The study design is a randomized double-blind randomized controlled trial.

Research Design

Patients will be randomly assigned to one of two treatment groups (see Intervention Description). Patients will randomly select one of 70 sealed envelopes the day of surgery. Patients will be blinded to the medication utilized as well as the treating surgeon (PI). A consecutive series of patients will be enrolled to prevent selection bias. A single surgeon will be performing all procedures to minimize variability. Upon completion of the surgery, a spinal needle will be loaded into the substance of the rotator cuff tendon under direct arthroscopic visualization. The surgeon will then leave the room and the envelope will be opened by the circulating operating room nurse. If the patient is in the treatment group, 2cc of an extracellular matrix graft be opened and then injected with a 22g spinal needle already placed into the bed of the repair by the physician assistant. Those patients that are in the control group will have the needle removed and no injection administered. The envelope will be then sealed with the patient's name and treatment group to allow for data analysis upon completion of the study.

Data Collection will occur post-operatively for 6 months. Data will be collected at 13 timepoints, in total for pain and opioid consumption. For the first seven days, data will be collected at 24-hour time intervals beginning the first morning after the surgery (POD1) at 8am then at 24-hour intervals for the next 7 days (POD7). Data will be collected using Oberd, an application that uses text message or email to collect information. The morning after the surgery (POD0) the first email will occur at 8am. Patients will then be notified by email alert 1 times per day (8am) asking to rate their pain on a scale of 0-10 (VAS) beginning on POD 1 thru POD 7. Patients will also respond to the number of pain pills taken in the slotted time span. All patients will be prescribed the same narcotic regimen (oxycodone IR) barring any allergies encountered. Patients who fail to respond to the email alert will be notified by the data collection system and contacted via phone by study personnel. Patients lacking smartphone technology will all be notified via telephone and also asked to keep a personal log to capture the information needed.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 and older
2. Primary diagnosis of rotator cuff tear, labral tear or SLAP tear
3. Able to provide informed consent
4. Is willing and able to accept text messages

Exclusion Criteria:

1. Older than 55 years old.
2. Pregnancy.
3. Known narcotic or alcohol abuse (< 3 months)
4. Revision shoulder surgery
5. Current narcotic regimen or contract with pain management specialist

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2020-12-04 (Actual); Primary Completion 2021-11-07 (Actual); Study Completion 2021-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: brian l badman, MD, Principal Investigator — American Health Network
Locations (1):
- American Health Network, Avon, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Colvin AC, Egorova N, Harrison AK, Moskowitz A, Flatow EL. National trends in rotator cuff repair. J Bone Joint Surg Am. 2012 Feb 1;94(3):227-33. doi: 10.2106/JBJS.J.00739. PMID 22298054
- [Background] Duellman TJ, Gaffigan C, Milbrandt JC, Allan DG. Multi-modal, pre-emptive analgesia decreases the length of hospital stay following total joint arthroplasty. Orthopedics. 2009 Mar;32(3):167. PMID 19309064
- [Background] Parvataneni HK, Shah VP, Howard H, Cole N, Ranawat AS, Ranawat CS. Controlling pain after total hip and knee arthroplasty using a multimodal protocol with local periarticular injections: a prospective randomized study. J Arthroplasty. 2007 Sep;22(6 Suppl 2):33-8. doi: 10.1016/j.arth.2007.03.034. Epub 2007 Jul 26. PMID 17823012

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1 participant was excluded after enrollment before assignment to a group because the participant did not meet age inclusion/exclusion criteria. 9 participants were enrolled but excluded from the study before assignment to groups because technical errors in data collection were identified before assignment.
Period: Overall Study
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft
Started | 5 | 0
Completed | 0 | 0
Not Completed | 5 | 0
Not completed — Participant outcomes data not collected due to technical errors. | 5 | 0

BASELINE CHARACTERISTICS:
Population: This study was halted due to failure of data collection system and first five randomized were all to control based on randomization.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft | Total
Number analyzed (Participants) | 5 | 0 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 0 | 5
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 5 | 0 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 0 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 4 | 0 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 5 |  | 5

OUTCOME MEASURES:

1. Primary Outcome: Patient Reported Post Operative Opioid Use
Description: Utilizing a prospective randomized controlled trial, narcotic use will be measured for 24-hour increments for a total of 7 post-operative days (PODs) then once on POD 14, 21, 28, and 42. Consumption will be measured by the number of tablets ingested and converted to morphine equivalent units and compared between the two treatment groups
Time Frame: Up till 6 weeks
Population: Due to technical errors in the participant-reported data collection system, no outcome measure data was collected from participants.
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Patient Reported Postoperative Pain: Visual Analogue Pain
Description: Utilizing a prospective randomized controlled trial, post-operative patient-reported VAS pain (on a scale of 0-10) will be collected 1 time per day (every 24 hours) for 7 post-operative days (PODs); then an average score collected on POD 14, POD 21, POD 28, and POD 42. Scores will be averaged and compared between the two treatment groups for the first 7 days, 2 week, 3rd week, 4th week and 6th week postoperatively. A score of zero will indicate no pain and a score of 10 will indicated maximum pain.
Time Frame: Up till 6 weeks
Population: as for outcome 1
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: American Shoulder and Elbow Scores
Description: To determine if there is a difference in American Shoulder and Elbow scores of patients with rotator cuff tears treated with and without the the ECM implant measured at 2 weeks, 6 weeks, 3 months and 6 months postoperatively. The scoring system is from 0 to a maximum of 100 with the higher scores indicating better outcomes.
Time Frame: Up till 6 months
Population: as for outcome 1
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft
Number analyzed (Participants) | 0 | 0

4. Other Pre Specified Outcome: Patient Reported Single Assessment Numeric Evaluation (SANE) Score
Description: Patient reported single assessment numeric evaluation (SANE) score (on a scale of 0 to 100%), measured preoperatively and postoperatively will be assessed for a difference; Scores will be checked at 2 weeks, 6 weeks, 3 months, and 6 months after surgery. A lower number indicates a poorer outcome and a higher number indicates a better outcome.
Time Frame: Up till 6 months
Population: as for outcome 1
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Shoulder Range of Motion
Description: Patients range of motion including forward flexion, abduction and external rotation will be measured preopertively and postoperatively with a manual goniometer at 6 weeks, 3 months, and 6 months postoperatively.
Time Frame: Up till 6 months
Population: as for outcome 1
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 11 months
Description: There were no adverse events to report for the 5 patients. All were control and no intervention. There were no serious adverse events for the five subjects.
Arm/Group | Group 1 Control | Group 2: ECM Injectable Graft
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/0
Other Adverse Events (participants affected / at risk) | 0/5 | 0/0

LIMITATIONS AND CAVEATS:
Trial terminated early because of technical problems with participant-reported data collection system. No outcome measure data was collected from participants. Once technical problems were identified and determined to be irreparable, the trial was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-10-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT04633837/Prot_SAP_000.pdf
  • Informed Consent Form (2020-12-04): https://cdn.clinicaltrials.gov/large-docs/37/NCT04633837/ICF_001.pdf